CLINICAL TRIAL: NCT02929082
Title: Interest of elastoFRM With Force Measure by MRI on Patients With Hepatocellular Cancer
Acronym: FORCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P150412
Record Dates: First submitted 2016-09-14; First posted 2016-10-10 (Estimated); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Hepatocellular Cancer
Keywords: magnetic resonance force
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 : volunteer patient (Experimental): Group 1 will be constituted of 20 volunteer patients coming for abdominal MRI with no known hepatic disease, in order to determine the feasibility of FRM . A 5-minute- additional sequence to measure FRM will be done for the volunteers.
  Interventions: Radiation: IRM with a 5-minute- additional sequence to measure FRM
- Group 2 : patient with resectable HCC (Experimental): Group 2 will be constituted of 60 patients with resectable HCC eligible for surgery. This group will enable to evaluate the gold standard.
  A 5-minute- additional sequence to measure FRM will be done while MRI sequence.
  Interventions: Radiation: IRM with a 5-minute- additional sequence to measure FRM
- Group 3 : patient with HCC eligible for TACE (Experimental): Group 3 will be constituted of 50 patients with HCC eligible for transplant with transcatheter arterial chemoembolization (TACE) treatment as pending treatment before transplant. This groups will enable to evaluate the efficiency of TACE through the necrosis percentage in treated HCC.
  A 5-minute- additional sequence to measure FRM will be done while MRI sequence
  Interventions: Radiation: IRM with a 5-minute- additional sequence to measure FRM

INTERVENTIONS:
Radiation: IRM with a 5-minute- additional sequence to measure FRM — IRM with a 5-minute- additional sequence to measure FRM for patients in group 1,2 and 3
  Other Names: FRM

SUMMARY:
FORCE project aims to measure actives forces of malignant tumor by magnetic resonance force (FRM). Two main forces are considered as key indicators of therapeutic response and metastatic potential: interstitial force and traction force at the interface cell/tumor. Biomarkers of these forces will be developped using direct images of magnetic resonance force (FRM). Efficiency of these non-invasive biomarkers will be evaluated through their capacity to predict tumoral environment invasion, notably micro-vascular invasion, and therapeutical results in Hepatocellular Cancer (HCC).

Principal criteria will be

1. micro-vascular invasion assessed by pathological examination of surgical pieces (gold standard).
2. interstitial force and traction force at the cell/tumor interface assessed by FRM.

Population of patients will be divided in three groups. A first group will be constituted of 20 volunteer patients coming for abdominal MRI with no known hepatic disease, in order to determine the feasibility of FRM. A second group will be constituted of 60 patients with resectable HCC eligible for surgery. This group will enable to evaluate the tumoral environment invasion. Third group will be constituted of 50 patients with HCC eligible for transplant with transcatheter arterial chemoembolization (TACE) treatment as pending treatment before transplant. This groups will enable to evaluate the efficiency of TACE through the necrosis percentage in treated HCC.

Inclusion of patients will occur during 24 months for a total study duration of 36 months.

All patients will have MRI as usual care. FRM is performed during MRI with the use of a specific medical device and therefore corresponds to an additional procedure of the research.

Moreover, patients in group 2 and 3 will be asked to participate to an ancillary study consisting in circulating tumoral cells (CTC) measurement. If they accept, a blood sample will be collected just before the MRI in order to evaluate the correlation between CTC and micro-vascular invasion.

DETAILED DESCRIPTION:
FORCE project aims to measure actives forces of malignant tumor by FRM. Two main forces are considered as key indicators of therapeutic response and metastatic potential: interstitial force and traction force at the cell/tumor interface. Biomarkers of these forces will be developped using direct images of magnetic resonance force (FRM). Efficiency of these non-invasive biomarkers will be evaluated through their capacity to predict tumoral environment invasion, notably micro-vascular invasion, and therapeutical results in Hepatocellular Cancer (HCC).

Principal criteria will be

1. micro-vascular invasion assessed by pathological examination of surgical pieces (gold standard).
2. interstitial force and traction force at the cell/tumor interface assessed by FRM.

Secondary criteria will be :

1. Percentage of nodular necrosis in HCC as a marker of a therapeutic response assessed by pathological examination of explant liver (gold standard).
2. interstitial force and traction force at the cell/tumor interface assessed by FRM.

Population of patients will be divided in three groups (see below). Inclusion of patients will occur during 24 months for a total study duration of 36 months.

Moreover, patients in group 2 and 3 will be asked to participate to an ancillary study consisting in circulating tumoral cells (CTC) measurement. If they accept, a blood sample will be collected just before the MRI in order to evaluate the correlation between CTC and micro-vascular invasion.

* Group 1 will be constituted of 20 volunteer patients coming for abdominal MRI with no known hepatic disease, in order to determine the feasibility of FRM.
* Group 2 will be constituted of 60 patients with resectable HCC eligible for surgery. This group will enable to evaluate the tumoral environment invasion. Patients of this group will be selected during multidisciplinary medical meetings. If they accept to participate to the ancillary study, a blood sample will be collected (2 tubes of 6 mL and 10 mL respectively) just before the MRI, an exam always performed before hepatic resection with a 5-minute- additional sequence to measure FRM. As soon as the surgery is performed, surgery pieces will be analysed by anatomopathology laboratory in order to assess, notably, presence of mirco-vascular invasion.
* Group 3 will be constituted of 50 patients with HCC eligible for transplant with transcatheter arterial chemoembolization (TACE) treatment as pending treatment before transplant. This groups will enable to evaluate the efficiency of TACE through the necrosis percentage in treated HCC. Patients of this group will be selected during multidisciplinary medical meetings. If TACE was already performed at inclusion and if patient accepts to participate to the ancillary study, a blood sample will be collected (2 tubes of 6 mL and 10 mL respectively) just before the MRI, an exam always performed before hepatic transplant with a 5-minute- additional sequence to measure FRM. As soon as the transplant is performed, surgery pieces (whole patient liver) will be analysed by anatomopathology laboratory in order to assess, notably, presence of necrosis on HCC nodules previously treated by TACE. If TACE was not performed at inclusion, TACE will be planified as usually. Data from TACE will be collected in the case report form (CRF). After TACE, same exams will be performed as described above.

All patients will have MRI as usual care. FRM is performed during MRI with the use of a specific medical device and therefore corresponds to an additional procedure of the research.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 : adults (≥ 18 y.o.) with life expectancy upper than 3 months; planified pancreatic or biliary MRI; signed informed consent form; affiliated to social security or equivalent.
* Group 2 : adults (≥ 18 y.o.) with life expectancy upper than 3 months; with HCC diagnosed by histological or cytological means or following EORTC/EASL criteria; eligible for HCC resection; treatment-naive patients for studied HCC lesion; signed informed consent form; affiliated to social security or equivalent.
* Group 3 : adults (≥ 18 y.o.) with life expectancy upper than 3 months; with HCC diagnosed by histological or cytological means or following EORTC/EASL criteria; eligible for hepatic transplant; eligible TACE treatment as pending treatment before transplant; treatment-naive patients for studied HCC lesion for treatments other than TACE; signed informed consent form; affiliated to social security or equivalent.

Exclusion Criteria:

* Group 1 : known chronic hepatic disease; contraindication for MRI as defined by the French Radiology Society.
* Group 2 : patients previously treated for studied HCC lesion; contraindication for MRI as defined by the French Radiology Society.
* Group 3 :patients previously treated for studied HCC lesion (except if TACE); contraindication for MRI as defined by the French Radiology Society.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Tumoral environment invasion assessed by the presence of microvascular invasion of the tumor capsule after pathological examination of the surgical pieces | 12 months

SECONDARY OUTCOMES:
therapeutical results of TACE assessed by percentage of nodular necrosis in HCC after pathological examination of the explant liver | 12 months
Interstitial force and traction force at the cell/tumor interface assessed by FRM | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Vilgrain, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Valérie Vilgrain, Clichy, France

IPD SHARING:
Plan to Share IPD: Undecided